CLINICAL TRIAL: NCT02692456
Title: Efficacy of Patient Position After Computerized Tomography Guided Antero-crural Celiac Trunk Neurolysis on Upper Abdominal Malignancy Pain
Brief Title: Effect of Patient Position on Computerized Tomography Guided Celiac Trunk Neurolysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: R,∕ 15.07.07
Record Dates: First submitted 2016-02-05; First posted 2016-02-26 (Estimated); Last update posted 2016-02-26 (Estimated); Status verified 2016-02

CONDITIONS: Upper Abdominal Malignancy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Double needle celiac neurolysis (DNCN) (Active Comparator): Patients were subjected to CT guided celiac neurolysis using 2 needle antero-crural technique on each side with patient in prone position and both needles will be lateral to the aorta
  Interventions: Device: Double needle celiac neurolysis (DNCN)
- Single needle celiac neurolysis (SNCN) (Placebo Comparator): Patients were subjected to CT guided celiac neurolysis using a single needle antero-crural approach from left side to be just in the front of the aorta near the origin of celiac trunk with patient in lateral position with his left side up then after the injection the patient were kept to his right side up for more homogenous spread of the dye.
  Interventions: Device: Single needle celiac neurolysis (SNCN)

INTERVENTIONS:
Device: Double needle celiac neurolysis (DNCN) — CT guided celiac neurolysis will be performed using 2 needles inserted on each sides of aorta where patient was positioned in prone position
  Arms: Double needle celiac neurolysis (DNCN)
Device: Single needle celiac neurolysis (SNCN) — CT guided celiac neurolysis will be performed through advancing a single needle to justfront of the aorta near the origin of celiac trunk where patient placed in lateral position
  Arms: Single needle celiac neurolysis (SNCN)

SUMMARY:
Computerized tomography-guided Celiac plexus neurolysis has become a popular technique. As, it has Cross-section imaging system to avoids anatomic structures injury, it has high density resolution that clearly display the retro-peritoneal anatomic structures ,it allow an optimal puncture site selection and measured the angle and depth of the needle insertion accurately with display the range of the neurolytic agent diffusion

DETAILED DESCRIPTION:
The aim of this study was to evaluate analgesic efficacy of a computerized tomography guided left lateral antero-crural approach near the origin of celiac trunk with patients position on their right side immediately after the procedure using a single needle injection technique for upper abdominal malignancy compared with the classic 2 needle posterior antero-crural injection technique and possible complications.

All patients will take thin computerized tomography section in the axial plane to detect the site of celiac plexus and coronal plane for correct site for needle placement.

Computerized tomography slices thickness will be from 3 mm at 5mm interval through all the abdominal and lower thoracic area. The celiac and superior mesenteric arteries will be identified after contrast injection.

When an ideal needle position and tip were confirmed, the stylet was removed and aspiration was performed to ensure that there was no blood is withdrawn.

A volume of 3 ml of lidocaine mixed with contrast was injected to confirm the position, after injection another cut has been taken to show the spread of contrast freely in the retro-peritoneal space around the celiac plexus and the aorta. After confirmation, that contrast was injected to surround the artery and make sure that there was no dorsal spread to avoid injury to somatic nerves. Also to make sure that there was no spread to the renal pelvis , injection of phenol 10% mixed with contrast through needle

ELIGIBILITY:
Inclusion Criteria:

* Patients with gastric carcinoma
* Patients with hepato-biliary-pancreatic cancer
* Patients with colonic malignancy
* Patients with peritoneal metastasis
* Patients with extensive hepatic metastasis
* Patients having intractable pain to opioids and other analgesics.
* Patients experienced adverse effects to opioids or other analgesics.
* Patients experienced improved intractable pain after diagnostic celiac plexus block

Exclusion Criteria:

* Patient's refusal
* Patients with bleeding tendency
* Patients with coagulopathy
* Patients who were benefited from oral analgesics with no serious side effects
* Patients with significant cardiac diseases
* Patients with organ failure
* Patients with distant vertebral metastasis
* Evidence of local infection at the puncture site
* Patients who did not experience improved pain after receiving a diagnostic celiac plexus block

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2015-06; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Failure rate of patients positioning | For 5 min before needle insertion
  Positioning failure means failure to put patient in prone or lateral position

SECONDARY OUTCOMES:
Time to achieve analgesia | for one hour after performing the procedure
  Time to achieve pain score less than 3
Failure of block | For 1 week after performing the procedure
  Failure of block is defined as patient having pain visual analogue scale greater than 3

CONTACTS AND LOCATIONS:
Overall Officials: Alaa A Elmaadawy, MD, Study Director — Lecturer of Anesthesia and Surgical Intensive Care; Ghada F EL-Rahmawy, MD, Principal Investigator — Professor of Anesthesia and Surgical Intensive Care; Nevert A Abdelghaffar, MD, Study Chair — lecturer of Anesthesia and Surgical Intensive Care
Locations (1):
- Mansoura University Cancer Institute, Al Mansurah, DK, Egypt

IPD SHARING:
Plan to Share IPD: Undecided